CLINICAL TRIAL: NCT05623566
Title: Evaluation of a Smartphone Based Screening Tool for Neonatal Jaundice in Surabaya, Indonesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After data quality check, inclusion criteria were not satisfied and data quality was poor. We concluded that results are not reliable
Sponsor: Picterus AS (Industry)
Collaborators: RSIA Kendangsaru Surabaya (Unknown); Universitas Airlangga (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/1608Indonesia
Record Dates: First submitted 2022-11-10; First posted 2022-11-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Experimental): In this study we aim to collect data of newborns with wider range of bilirubin levels to adjust the Picterus JP algorithm and optimize the app performance. This will enable a high qualitative estimation of bilirubin levels in the blood of new-borns for all skin colors.
  Interventions: Device: Picterus Jaundice Pro

INTERVENTIONS:
Device: Picterus Jaundice Pro — In this study we aim to collect data of newborns with wider range of bilirubin levels to adjust the Picterus JP algorithm and optimize the app performance. This will enable a high qualitative estimation of bilirubin levels in the blood of new-borns for all skin colors.
  Other Names: Picterus JP

SUMMARY:
A cross-sectional conductive study aiming to evaluate the accuracy of a novel smartphone application that estimates bilirubin levels in newborns in Surabaya.

DETAILED DESCRIPTION:
A cross-sectional conductive study aiming to evaluate the accuracy of a novel smartphone application that estimates bilirubin levels in newborns at Airlangga University hospital and RSIA Kendangsari MERR in Surabaya.

This cross-sectional study evaluates the accuracy of a novel smartphone application that estimates bilirubin levels in Indonesian newborns. The Picterus Calibration Card was placed on the chest of the newborn with the hole in the card placed over the infant's sternum. A validated smartphone with Picterus JP was used to collect digital images.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with gestational age >31
* Birth weight ≥ 1500g
* Age 0 - ≤14 days
* Consent obtained from the parents

Exclusion Criteria:

* Infants born with congenital abnormalities;
* Infants respiratory support;
* Infants suffering from a condition that may alter the skin tissue circulatory system, such as sepsis and heart failure;
* Infants who have received phototherapy in the last 24 hours.

Ages: 1 Hour to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of newborns, independent of skin color, using Picterus JP. | 5-10 minutes
  Evaluate of smartphone-based screening tool (Picterus JP) for neonatal jaundice in Indonesian newborns.

SECONDARY OUTCOMES:
Correlation between bilirubin estimates in from a smartphone application and bilirubin measurements in serum in newborn | 1-2 minutes
  To evaluate the correlation between bilirubin estimates in from a smartphone application and bilirubin measurements in serum in newborns with varying degree of jaundice
correlation between bilirubin estimates from a smartphone application and bilirubin estimates from a standard transcutaneous device in newborns | 5-10 minutes
  To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from a standard transcutaneous device in newborns with varying degree of jaundice
Correlation between bilirubin estimates from a smartphone application and bilirubin estimates from visual inspection in newborns | 5-10 minutes
  To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from visual inspection in newborns with varying degree of jaundice

CONTACTS AND LOCATIONS:
Locations (3):
- Indonesia (3):
  - Airlangga University hospital, Surabaya, East Java
  - RSIA Kendangsari MERR, Surabaya, East Java
  - Dr. Soetomo General Hospital, Surabaya, East Java